CLINICAL TRIAL: NCT04230733
Title: Correlation Analysis of Pelvis Displacement and Gait Indicators in Patient With Lumbar Disc Herniation : Retrospective Study Using Electronic Medical Record Data
Brief Title: Pelvis Displacement and Gait Indicators in Patient With Lumbar Disc Herniation
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2018-08
Record Dates: First submitted 2019-11-13; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-11

CONDITIONS: Lumbar Disc Herniation; Gait Analysis; Pelvis Abnormal
Keywords: Gait; Pelvic height; Leg Length Discrepancy; Sacral angle
MeSH Terms: conditions — Intervertebral Disc Displacement; Leg Length Inequality

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate the correlation between pattern of gait and pelvic displacement in patients with lumbar disc herniation.

DETAILED DESCRIPTION:
Walking is a repetitive movement that moves your body while keeping your posture stable. The pelvis is located between the hip and lumbar region, where many muscles are attached to regulate the movement of the hip and lumbar spine. Asymmetrical pelvic alignment affects stability of the lower extremities and trunk, making normal walking difficult. The purpose of this study is to investigate the pattern of gait according to pelvic displacement in patients with lumbar disc herniation.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar intervertebral disc herniation as confirmed by a doctor of medicine or a doctor of Korean medicine through an MRI
* Patient who got gait analysis

Exclusion Criteria:

* Patients without MRI and X-ray
* Patient diagnosed with ankle disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted to Jaseng Hospital of Korean Medicine and got gait analysis
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Correlation between pelvic displacement and gait parameters | A week after data collected
  <Pelvic displacement>
  * Sacral angle : The angle between the parallel line drawn on the first vertebral body(Sacrum) and the horizontal line
  * Leg Length Discrepancy : Difference between the values of both sides by measuring the height of the upper edge of both femoral heads
  * Pelvic height : Difference between the left and right peaks of both iliac crests
  * Gravity line : Line passing through the gravity point(L3) of the human body
  <Gait parameters>
  Step, Stance phase, Swing phase, Single support, Double support, Step time, Stride, Cadence, Load response, Pre swing, Gait cycle, Speed, Acceleration, contact phase, foot flat, propulsive, PCI

SECONDARY OUTCOMES:
Numeric Rating Scale | A week after data collected
  Using NRS-11(0 to 10) which is measured at first visit

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, KMD, Ph.D, Study Director — Jaseng Medical Foundation
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No